CLINICAL TRIAL: NCT05490069
Title: The Effect of Instant Message Intervention for Psychological Well-being Among Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-526
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Depressive Symptoms; Mobile Phone Use
MeSH Terms: conditions — Stroke; Depression; Cell Phone Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receive iCBT based EMI with message content, delivery frequency and timing personalised to participants' preferences.
  Interventions: Other: iCBT-based EMI
- Control group (No Intervention): Receive general mental health information through instant message.

INTERVENTIONS:
Other: iCBT-based EMI — Consists of brief iCBT for psychological support (mandatory), stroke care education (optional), and real-time chat-based support messages, delivered according to participants' preferences.
  Arms: Intervention group

SUMMARY:
The proposed pilot trial aims to evaluate the feasibility of iCBT based EMI, which is a real-time, real-world, personalised and cost-effective approach, for stroke survivors' psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke (ICD-10 codes: I60-I69)
* Aged ≥18
* Able to read and communicate in Chinese (Cantonese or Putonghua)
* Able to use text messaging function on mobile phones
* MoCA 5-minute Protocol (cognitive screen) ≥14 (Equivalence to MMSE ≥ 21)
* Discharged home from hospital within preceding 6 months
* PHQ-9 (depressive symptom) score range from 5 to 19 (cf. mild: 5-9, moderate: 10-14, moderately severe: 15-19 and severe: 20-27)

Exclusion Criteria:

* Currently receiving active stroke care in acute or post-acute inpatient settings
* Has diagnosis of psychiatric disease or is currently taking psychotropic drug
* PHQ-9 ≥ 20 (i.e., severe depressive symptom)
* Currently participating in any type of psychological intervention (e.g., CBT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (Patient Health Questionnaire-9 [PHQ-9]) | 24-week
  A 9-item scale with score ranging from 0 to 27, higher scores indicate higher severity of depressive symptom

SECONDARY OUTCOMES:
Anxiety symptoms (Generalized Anxiety Disorder-7 [GAD-7]) | 24-week
  A 7-item scale with score ranging from 0 to 21, higher scores indicate higher severity of anxiety symptoms
Stress level (Perceived Stress Scale [PSS-4]) | 24-week
  A 4-item scale with score ranging from 0 to 16, higher scores indicate higher severity of stress
Spiritual well-being (Sub-scale of Spirituality Scale for Chinese Elders [SSCE]) | 24-week
  An 8-item scale with score ranging from 0 to 32, higher scores indicate better spiritual well-being
Loneliness (UCLA Loneliness Scale [ULS-8]) | 24-week
  An 8-item scale with score ranging from 8 to 32, higher scores indicate higher level of loneliness

CONTACTS AND LOCATIONS:
Locations (7):
- Hong Kong (7):
  - Hong Kong PHAB Association, Hong Kong
  - Hong Kong Stroke Association, Hong Kong
  - NT West Community Rehabilitation Day Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Hong Kong Society for Rehabilitation, Hong Kong
  - Tung Wah Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No